CLINICAL TRIAL: NCT06289725
Title: Impact of Hepatitis B Virus Genotype on Treatment Response in Children With Chronic Hepatitis B
Status: Recruiting | Type: Observational
Sponsor: Ly Hoa Anh Minh (Other)
Responsible Party: Sponsor-Investigator, Ly Hoa Anh Minh, PhD student, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: IRB-VN01002-23932
Record Dates: First submitted 2024-02-24; First posted 2024-03-04 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis b
Keywords: Hepatitis B; treatment response; genotype; children
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with genotype B
  Interventions: Drug: antiviral treatment
- patients with genotype C
  Interventions: Drug: antiviral treatment

INTERVENTIONS:
Drug: antiviral treatment — The patient was treated with antiviral drugs according to the protocol of the Ministry of Health of Vietnam 2019

SUMMARY:
The study aimed to evaluate the relationship between hepatitis B virus genotype and treatment response in children with chronic hepatitis B with specific treatment indications. This is a prospective cohort study, with a follow-up period of at least 12 months, conducted at Children's Hospital 1 and City Children's Hospital, Ho Chi Minh City, Vietnam. The patient's blood was taken to be tested for hepatitis B virus genotyping using Sanger sequencing at the Center for Molecular Biomedicine Ho Chi Minh City. The research hypothesis is that genotype is related to treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 years old to under 16 years old are diagnosed with hepatitis B chronic disease AND
* HBsAg or HBV DNA: positive for at least six months AND
* Liver enzyme ALT: continuously increased by> 70 for male and > 50 for female (> 2 x ULN) AND
* The virus is proliferating: HBV DNA above 20,000 IU/mL (if HBeAg positive) OR HBV DNA above 2,000 IU/mL (if HBeAg negative) AND
* A parent or legal guardian of the pediatric patient obtains consent for them to participate in research.

Exclusion Criteria:

* HIV and hepatitis C co-infection
* Patients have other chronic liver disease (Wilson, autoimmune hepatitis)
* Patients are being treated with immunosuppressive drugs
* Psychomotor retardation, cerebral palsy, brain sequelae

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with chronic hepatitis B are indicated for drug treatment antiviral treatment at Children's Hospital 1 and City Children's Hospital, Ho Chi Minh City, Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Serological response for HBeAg | 12 months after treatment
  Serological response for HBeAg applies only to patients with HBeAg-positive Chronic Hepatitis B and is defined as HBeAg loss and seroconversion to anti-HBe.

SECONDARY OUTCOMES:
Virological response | 12 months after treatment
  Virological response is defined as undetectable HBV DNA by a sensitive PCR assay.

OTHER OUTCOMES:
Biochemical response | 12 months after treatment
  Biochemical response is defined as normalisation of ALT levels

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Children's Hospital 1, Ho Chi Minh City
  - City Children's Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KJ, Choe BH, Choe JY, Kim JY, Jeong IS, Kim JW, Yang HR, Chang JY, Kim KM, Moon JS, Ko JS. A Multicenter Study of the Antiviral Efficacy of Entecavir Monotherapy Compared to Lamivudine Monotherapy in Children with Nucleos(t)ide-naive Chronic Hepatitis B. J Korean Med Sci. 2018 Feb 19;33(8):e63. doi: 10.3346/jkms.2018.33.e63. PMID 29441755
- [Result] Kao JH, Chen PJ, Lai MY, Chen DS. Hepatitis B virus genotypes and spontaneous hepatitis B e antigen seroconversion in Taiwanese hepatitis B carriers. J Med Virol. 2004 Mar;72(3):363-9. doi: 10.1002/jmv.10534. PMID 14748059
- [Result] Chien RN, Yeh CT, Tsai SL, Chu CM, Liaw YF. Determinants for sustained HBeAg response to lamivudine therapy. Hepatology. 2003 Nov;38(5):1267-73. doi: 10.1053/jhep.2003.50458. PMID 14578866